CLINICAL TRIAL: NCT03779815
Title: A Pilot Phase 2, Open-label, Non-randomized, Single Center Study to Explore Diagnostic Validity of [18F]Florbetaben Positron Emission Tomography for Detecting Amyloidosis in Multiple Myeloma Patients
Brief Title: Detection of Amyloidosis in Multiple Myeloma Patients by [18F]Florbetaben Positron Emission Tomography
Acronym: PET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ulsan University Hospital (Other)
Responsible Party: Principal Investigator, Jae-Cheol Jo, Assistant professor, Ulsan University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: UUH-2018-05-034-001
Record Dates: First submitted 2018-09-12; First posted 2018-12-19 (Actual); Last update posted 2019-04-18 (Actual); Status verified 2019-04

CONDITIONS: Multiple Myeloma
Keywords: multiple myeloma; amyloidosis; Florbetaben
MeSH Terms: conditions — Multiple Myeloma; Amyloidosis | interventions — 4-(N-methylamino)-4'-(2-(2-(2-fluoroethoxy)ethoxy)ethoxy)stilbene

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- [18F]Florbetaben PET/CT imaging (Experimental): * Maximally 18 subjects with multiple myeloma (up to 6 subjects in whom amyloidosis in suspected and up to 12 subjects in whom amyloidosis is not suspected)
  * Intravenous injection of [18F]Florbetaben and PET/CT scanning
  * Intervention: Drug ([18F]Florbetaben)
  Interventions: Drug: [18F]Florbetaben

INTERVENTIONS:
Drug: [18F]Florbetaben — * Drug: [18F]Florbetaben
  * [18F]Florbetaben PET/CT Imaging for detecting amyloidosis in multiple myeloma
  * Other name: Neuraceq
  * Amount: 300 MBq ± 20% bolus, 10mL intravenously
  Other Names: neuraceq

SUMMARY:
[18F]Florbetaben PET/CT imaging will noninvasively assess amyloid deposition in systemic amyloidosis.

DETAILED DESCRIPTION:
Diagnostic validity of [18F]Florbetaben PET for detecting amyloidosis will be assessed in subjects with multiple myeloma.

ELIGIBILITY:
Inclusion Criteria:

* Subject is over 19 years old and male or female of any race/ethnicity
* Subject has been diagnosed with multiple myeloma by a hemato-oncology specialist
* Subject has undergone clinical, laboratory, or imaging work-up if amyloidosis is suspected
* Subject has voluntarily agreed to participate in the study

Exclusion Criteria:

* Subject or subject's legally acceptable representative does not provide written informed consent.
* Female subject is pregnant or nursing. Exclusion of the possibility of pregnancy is made by one of the following: 1) Woman is physiologically post-menopausal (cessation of menses for more than 2 years), 2) woman is surgically sterile (has had a documented bilateral oophorectomy and/or documented hysterectomy, or 3) if the woman is of childbearing potential, a serum or urine pregnancy test performed within 24 hours immediately prior to administration of [18F]Florbetaben has to be negative and the women is advised to apply contraceptive measures during her participation in this study.
* Subject has concurrent severe and/or uncontrolled and/or unstable medical disease (which could compromise participation in the study) in the judgment of the investigator.
* Subject has received any investigational drugs or devices within four weeks prior to the study enrollment.
* Subject has been previously included in this study.
* Subject has any other condition or personal circumstances that, in the judgment of the investigator, might make collection of complete data difficult or impossible.
* Subject is allergic to Florbetaben or any of ingredients of Florbetaben

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2018-08-20 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2019-02-28 (Actual)

PRIMARY OUTCOMES:
sensitivity and specificity per patient analysis | Up to 6 months after [18F]Florbetaben PET/CT scanning
  Sensitivity and specificity of [18F]Florbetaben PET/CT for the diagnosis of subjects with clinical, laboratory, radiological, or histopathological evidence of amyloidosis

SECONDARY OUTCOMES:
sensitivity and specificity per organ analysis | Up to 6 months after [18F]Florbetaben PET/CT scanning
  Sensitivity and specificity of [18F]Florbetaben PET/CT for the diagnosis of affected organs with clinical, laboratory, radiological, or histopathological evidence of amyloidosis
Correlation with severity | Up to 6 months after [18F]Florbetaben PET/CT scanning
  Correlation of [18F]Florbetaben activity with clinical/radiological/histopathological indices of amyloidosis severity
Adverse events | Up to 28 days after [18F]Florbetaben PET/CT scanning
  Adverse events will be monitored.

CONTACTS AND LOCATIONS:
Overall Officials: Jae-Cheol Jo, PhD, Principal Investigator — Ulsan University Hospital
Locations (1):
- Ulsan University Hospital, Ulsan, South Korea

IPD SHARING:
Plan to Share IPD: No